CLINICAL TRIAL: NCT04753424
Title: Autologous Semitendinosus Tendon Graft as Meniscal Transplant - a Clinical Pilot Study
Brief Title: Semitendinosus Graft as Meniscal Transplant
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Karl O. Eriksson, Associate Professor, Karolinska Institutet
Other Study IDs: semiTmeniscus
Record Dates: First submitted 2021-01-06; First posted 2021-02-15 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Patient Satisfaction; Graft Failure; Osteo Arthritis Knee; ACL; Meniscus Tear
Keywords: meniscus transplantation
MeSH Terms: conditions — Patient Satisfaction | interventions — Wound Closure Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgical technique — Description of novel surgical technique using autologous semitendinosus graft as meniscus transplant.

SUMMARY:
Removal of meniscal tissue is described to result in poor knee function and a significant risk for future development of osteoarthritis. Different implants have been suggested to substitute a removed meniscus. Meniscal allograft transplantation is not widely available due to costs and availability. The semitendinosus tendon is a known graft with biological properties with potential to remodel and revascularize in an intraarticular environment such as anterior cruciate ligament reconstruction. The objective for this study was to investigate whether the semitendinosus tendon graft could function as a meniscal transplant.

ELIGIBILITY:
Inclusion Criteria:

* Previous subtotal or total meniscectomy
* Post meniscectomy symptoms
* No osteoarthritic changes on radiography more than Ahlbäck 1
* Knee aligment (hip-knee-angle) +/- 3°
* No persisting ACL insufficiency

Exclusion Criteria:

* Difficulty understanding the instructions
* Current psychiatric diagnosis
* Smoking

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients, both male and female, 20-50 years of age, with previous subtotal or total meniscectomy, suffering from post meniscectomy symptoms are assessed at the outpatient clinic. If inclusion criteria are met, the patients receive information regarding the treatment.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Failure | 2 years
  Surgical failure of transplant defined as meniscus symptoms (joint line tenderness, swelling, locking or positive McMurray) resulting in a need for re-arthroscopy and subtotal or total resection of the transplant.

SECONDARY OUTCOMES:
Improved subjective knee function | 2 years
  Patient reported outcome measure using the Knee Injury and Osteoarthritis Outcome Score (KOOS), 0-100 where 100 indicate best possible result.
Improved subjective knee function | 2 years
  Patient reported outcome measure using Lysholm (0-100 where 100 indicate best possible result) and Tegner activity score (0-10, where 10 indicate the highest activity level) .
Improved subjective knee function | 2 years
  Patient reported outcome measure using Euroqol 5 dimensions (EQ-5D) score (quality of life instrument with five dimensions with points from 1 to 3 where 1 indicates no problem and 3 indicate severe problems).
Improved subjective knee function | 2 years
  Patient reported outcome measure using Global score (0-10 where 10 indicate best possible result)

CONTACTS AND LOCATIONS:
Locations (1):
- KISÖS, Stockholm, Sweden

REFERENCES:
- [Background] Kohn D. Autograft meniscus replacement: experimental and clinical results. Knee Surg Sports Traumatol Arthrosc. 1993;1(2):123-5. doi: 10.1007/BF01565466. PMID 8536007
- [Background] Johnson LL, Feagin JA Jr. Autogenous tendon graft substitution for absent knee joint meniscus: a pilot study. Arthroscopy. 2000 Mar;16(2):191-6. doi: 10.1016/s0749-8063(00)90035-5. PMID 10705332
- [Background] Ayala Mejias JD, Sciamanna RC, Muniesa MP, Perez-Espana LA. A case report of semitendinosus tendon autograft for reconstruction of the meniscal wall supporting a collagen implant. BMC Sports Sci Med Rehabil. 2013 Mar 28;5:4. doi: 10.1186/2052-1847-5-4. PMID 23557091

DOCUMENTS (1):
  • Study Protocol (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT04753424/Prot_000.pdf